CLINICAL TRIAL: NCT03321188
Title: Heated Intraperitoneal Chemotherapy in Primary Ovarian Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrea Jewell (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor-Investigator, Andrea Jewell, Medical Doctor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2017-HIPEC-Ovarian
Record Dates: First submitted 2017-06-29; First posted 2017-10-25 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer
Keywords: Heated intraperitoneal chemotherapy; HIPEC; cisplatin; paclitaxel; carboplatin; adjuvant IV chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HIPEC + adjuvant IV chemotherapy (Experimental): HIPEC
  * HIPEC will be administered intraoperatively one time only.
    *HIPEC cisplatin will be administered at rate of 100 milligram per meter squared (mg/m2)
  * Administration of HIPEC will have a duration of 90 minutes.
  Adjuvant IV chemotherapy
  * IV Paclitaxel
    * Dose: 80mg/m2 IV over 1 hour
    * Schedule: Days 1, 8 and 15
    * Cycle Length: 3 weeks (21 days)
  * IV Carboplatin
    * Dose: Area under the curve (AUC) 6 IV
    * Schedule: Day 1
    * Cycle Length: 3 weeks (21 days)
  Interventions: Procedure: HIPEC; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Procedure: HIPEC — HIPEC with cisplatin
Drug: Carboplatin — Adjuvant IV chemotherapy
Drug: Paclitaxel — Adjuvant IV chemotherapy

SUMMARY:
This study will evaluate the use of Heated Intraperitoneal Chemotherapy (HIPEC) for primary treatment of ovarian cancer at the time of surgical debulking, to assess if intravenous (IV) chemotherapy can be started within 42 days of HIPEC and cytoreduction. All patients will receive cytoreductive surgery followed by a one-time closed HIPEC with cisplatin at 41-43 degrees Celsius for 90 minutes in the operating room. This is followed by 6 cycles of intravenous carboplatin and paclitaxel on an outpatient basis.

DETAILED DESCRIPTION:
Heated Intraperitoneal chemotherapy (HIPEC) has several potential benefits. High-dose chemotherapy can be used due to the plasma-peritoneal barrier resulting in little absorption into the blood stream. Additionally, there is higher peritoneal penetration in comparison to IV regimen, and does not have the limitation of traditional IP regimen of post-operative adhesions. Hyperthermia itself has cytotoxic effects and can increase the depth of tumor penetration by the chemotherapeutic agent up to 3 millimeters; moreover, hyperthermia can potentiate its antineoplastic effects.

In recent times, morbidity and mortality associated with HIPEC has drastically improved. One large retrospective review of 694 patients, treated between 2005 and 2011, utilizing the American College of Surgeons National Surgical Quality Improvement Program (ACS NSQUIP) database, demonstrated a complication rate of 33% and 30-day mortality of 2.3%, both rates consistent with outcomes for other major complex abdominal operations.

Recently, a Phase I dose escalation study to evaluate maximum tolerated dose (MTD) of HIPEC administration of cisplatin in recurrent epithelial ovarian cancer (EOC) patients was published. The MTD of cisplatin was 100 milligrams per meter squared (mg/m2) with no mortality or safety concerns. While the trial had only 12 patients, all were able to receive post-operative IV chemotherapy, with all patients completing at least five cycles.

In protocol Gynecologic Oncology Group (GOG)-0172, intraperitoneal cisplatin and paclitaxel, plus intravenous paclitaxel, demonstrated the longest median survival reported in optimally debulked stage III ovarian cancer. Currently, the GOG is studying variations of the intraperitoneal (IP) regimen to preserve the survival advantage, but make it tolerable for patients to receive 6 cycles without discontinuing therapy due to distress and toxicity. The importance of developing an acceptable GOG-0172 alternative is emphasized by the recent National Cancer Institute (NCI) Clinical Announcement recognizing the superiority of intraperitoneal chemotherapy in the optimal disease setting.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent.
* Patients with a histologic diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma, Stage 3(III)B - 3(III)C with optimal (≤ 1 centimeter) residual disease.
* Patients with the following histologic epithelial cell types are eligible:
* Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, or adenocarcinoma not otherwise specified.
* No previous HIPEC.
* Patient has a planned cytoreduction surgery - Note: registration occurs during surgery and not before; if, during surgery, the Principal Investigator/Sub-Investigator discerns that all disease cannot be removed surgically, the participant will be considered a "screen failure", HIPEC will not be performed, and the participant will be removed from the study.
* Age ≥ 18 years.
* Performance Status Eastern Cooperative Group (ECOG) 0- 2
* Adequate organ and marrow function as defined below:

  1. absolute neutrophil count ≥ 1.5 kilograms per microliter (K/UL)
  2. platelets ≥ 100 K / UL
  3. total bilirubin within 1.5 x normal institutional limits
  4. Aspartate Aminotransferase (AST) / Serum Glutamic Oxaloacetic Transaminase (SGOT) ≤ 2.5 X institutional upper limit of normal
  5. Alanine Aminotransferase (ALT) / Serum Glutamic Pyruvic Transaminase (SPGT) ≤ 2.5 X institutional upper limit of normal
  6. creatinine within 1.5 x normal institutional limits

     * Note: If a potential participant has non-clinically significant variances related to the organ and marrow parameters listed above, PI review and approval is required before enrollment.
* Women of child-bearing potential and their male partners also of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  *A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy; OR Has not been naturally postmenopausal for at least 12 consecutive months (has had menses at any time in the preceding 12 consecutive months)

  *Note: Acceptable forms of birth control are listed below:
* One Barrier method (cervical cap with spermicide plus male condom; diaphragm with spermicide plus male condom) Plus Hormonal method (oral contraceptives, implants, or injections) or an intrauterine device (e.g., Copper-T).

Exclusion Criteria:

Participants meeting any of the exclusion criteria listed below at screening will be excluded from study participation.

* Current or anticipated use of other investigational agents.
* Patient has received chemotherapy or radiotherapy within 4 weeks prior to entering the study or has not recovered sufficiently (PI will judge patient recovery status) from adverse events due to agents administered more than 4 weeks earlier.
* Patient has history of or currently has non-peritoneal surface macroscopic metastatic disease in addition to peritoneal surface malignancy such as macroscopic pulmonary disease or other macroscopic disease outside of the peritoneal cavity.
* Patients with a current diagnosis of borderline epithelial ovarian tumor (formerly "tumors of low malignant potential") or recurrent invasive epithelial ovarian cancer treated with surgery only (such as those with stage Ia or Ib low Grade lesions) are not eligible. Patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated, new invasive epithelial ovarian or peritoneal primary cancer are eligible, provided that they have not received prior chemotherapy for any ovarian tumor.
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: Stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other International Federation of Gynecology and Obstetrics (FIGO) Grade 3 lesions.
* ECOG 3 - 4
* Patients with history or current diagnosis of inflammatory bowel disease are not eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Cisplatin, carboplatin and paclitaxel or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Current psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to start of intravenous (IV) chemotherapy. | 42 days
  Time will be measured in days starting at the time of the completion of HIPEC surgery and ending at the time of initiation of chemotherapy.

SECONDARY OUTCOMES:
Chemotherapy-related adverse events. | 90 days
  Chemotherapy-related adverse events will be defined per the Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Proportion of deaths occurring in hospital. | Up to 2 years
  Assess using Participant Electronic Medical Record indicating time of death.
Proportion of deaths occurring during post-hospital discharge period. | 30 days
  Assess using Participant Electronic Medical Record indicating time of death.
Proportion of deaths occurring during post-hospital discharge. | 90 days
  Assess using Participant Electronic Medical Record indicating time of death.
Average number of days in hospital Intensive Care Unit (ICU). | Up to 2 years
  Assessed from the time of surgery until the transition out of ICU.
Average overall length of in-hospital stay. | Up to 2 years
  Defined as days from the time of admission for surgery until discharge date of initial hospitalization
Average number of hospital re-admissions. | 90 days
  Assessed from the time of initial hospitalization discharge date.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Jewell, MD, Principal Investigator — The University of Kansas - Cancer Center
Locations (1):
- The University of Kansas Cancer Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No